CLINICAL TRIAL: NCT03642821
Title: Intracranial Aneurysms Treatment With the OPTIMA Coil System
Acronym: INSTANT
Status: Completed | Type: Observational
Sponsor: Balt Extrusion (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP-201702-OPTIMA
Record Dates: First submitted 2018-08-10; First posted 2018-08-22 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Intracranial Aneurysm; Coiling Therapy
Keywords: coil; aneurysm
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: intracranial aneurysm coiling — endovascular treatment of intracranial aneurysm by coiling procedure using OPTIMA coils system
  Other Names: OPTIMA coils

SUMMARY:
International, non-randomized, European , multicenter, observational study to collect data for the treatment of intracranial aneurysms with OPTIMA coils system to further document its safety and efficacy

ELIGIBILITY:
Inclusion Criteria:

1. Patient with small or large intracranial aneurysm, ruptured or unruptured, intended to be selectively treated with the OPTIMA coil system. Patients with recanalized aneurysms previously treated with coils exclusively are also eligible. Balloon and stent assisted coiling are allowed at index procedure.
2. In case of multiple aneurysms, patient can be included when only 1 aneurysm is treated during the procedure and none of the other aneurysms are treated up to 30 days post-procedure
3. Patient older than 18 years
4. Patient who has been informed of the study and has signed an informed consent form where applicable according to local regulations.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. giant aneurysms (>25 mm)
  2. recanalized aneurysms initially treated with stent or flow diverter (Only aneurysms initially treated with coils are eligible)
  3. aneurysm treated with parent artery occlusion
  4. dissecting or fusiform aneurysms
  5. aneurysms associated with an arteriovenous malformation
  6. aneurysm intended to be treated with flow diverter or flow disrupter during the procedure
  7. aneurysm intended to be treated in a staged procedure
  8. intracranial tumor (except meningioma)
  9. Any condition or any situation that would prohibit the patient from coming to the investigational center for the follow-up, as requested according to sites current practice.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Morbi-mortality at 30 days | 30 days
  Rate of adverse events including thromboembolic events, the bleeding/rebleeding episodes, the rate of retreated aneurysm and the rate of mortality occurring during the procedure and up to 30 days.
Clinical outcomes (mRS) at 30 days | 30 days
  Classification of the patient clinical and neurological outcomes based on modified Rankin Scale from 0 (no symptoms a all) to 6 (dead). Global outcomes of mRS 0-2 are considered good and those of mRS 3-6 (including mRS 6 - deceased) are considered to be poor.

SECONDARY OUTCOMES:
Morbi-mortality at 12 months | 12 months
  Rate of adverse events including thromboembolic events, the bleeding/rebleeding episodes, the rate of retreated aneurysm and the rate of mortality occurring within 12 months after the procedure.
Clinical outcomes (mRS) at 12 months | 12 months
  Classification of the patient clinical and neurological outcomes based on modified Rankin Scale from 0 (no symptoms a all) to 6 (dead). Global outcomes of mRS 0-2 are considered good and those of mRS 3-6 (including mRS 6 - deceased) are considered to be poor.
Aneurysm occlusion rate | Up to 24h and 12 months
  Post-procedure and 12-month follow-up efficacy based on the assessment of the aneurysm occlusion rate according to the 3-grade Montreal scale (complete occlusion/neck remnant/aneurysm remnant).

CONTACTS AND LOCATIONS:
Locations (20):
- Medizinische Universität Innsbruck, Innsbruck, Austria
- France (9):
  - CHU de Bordeaux - Hôpital Pellegrin, Bordeaux
  - CHU de Brest - Hôpital La Cavale Blanche, Brest
  - Hospices Civils de Lyon - Hôpital Neurologique, Bron
  - CHU Côte de Nâcre, Caen
  - Hôpital Privé Clairval, Marseille
  - CHU Gui de Chaulliac, Montpellier
  - CHU Hôpital Maison Blanche, Reims
  - CHU Charles-Nicolle, Rouen
  - CHRU Strasbourg Hautepierre, Strasbourg
- Zentralklinikum Augsburg, Augsburg, Germany
- Italy (4):
  - Azienda Ospedallera, Catania
  - San Gerardo Hospital, Monza
  - Antonio Cardarelli Hospital, Napoli
  - ULSS8 Berica Ospedale San Bortolo, Vicenza
- University of Latvia, Faculty of Medicine, Riga, Latvia
- Spain (3):
  - Hospital Universitario de Burgos, Burgos
  - Hospital: Fundacion Jimenez Diaz, Madrid
  - Hospital: Puerta de Hierro, Madrid
- HUG Hôpital cantonal universitaire de geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No